CLINICAL TRIAL: NCT07069556
Title: ColoSense Post Approval Study
Brief Title: ColoSense Post-Approval Study
Status: Recruiting | Type: Observational
Sponsor: Geneoscopy, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-PRT-0004
Record Dates: First submitted 2025-06-27; First posted 2025-07-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer (Diagnosis)
MeSH Terms: conditions — Colorectal Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: ColoSense — multi-target stool RNA test

SUMMARY:
The post-approval study (PAS) described here will supplement existing data generated in the CRC-PREVENT clinical trial. The primary outcomes of this supplemental study will include: clinical sensitivity, clinical specificity, positive predictive value (PPV), and negative predictive value (NPV) of ColoSense.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, ≥45 years of age (subjects aged 18-45 can be enrolled onto the clinical trial but are not eligible for primary endpoint analysis)
* Subject is able to understand the study procedures, and is able to provide consent to participate in the study and authorizes release of relevant protected health information through reviewing and consenting to a HIPAA medical release form
* Subject is able and willing to provide stool samples within the 120 days prior to a colonoscopy procedure
* Subject is able and willing to undergo a colonoscopy after providing a stool sample

Exclusion Criteria:

* Subject had any precancerous findings on most recent colonoscopy. This does not include benign, and/or hyperplastic polyps of any size
* Subject has a history or diagnosis of colorectal cancer
* Subject has a history of aerodigestive tract cancer
* Subject has had a positive non-invasive screening diagnostic within the associated recommended intervals:

  * Fecal occult blood test or fecal immunochemical test within the previous twelve (12) months
  * FIT-DNA test within the previous 36 months
* Subject has had a colonoscopy in the previous nine (9) years.
* Subject has had a prior colorectal resection for any reason other than sigmoid diverticular disease
* Indication for colonoscopy was due to overt rectal bleeding, e.g., hematochezia or melena, within the previous 30 days. (Blood on toilet paper, after wiping, does not constitute rectal bleeding)
* Subject has a diagnosis or personal history of any of the following high-risk conditions for colorectal cancer:

  * Inflammatory bowel disease (IBD) including chronic ulcerative colitis (CUC) and Crohn's disease
  * Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP)
  * Hereditary non-polyposis colorectal cancer syndrome (also referred to as "HNPCC" of "Lynch Syndrome")
  * Other hereditary cancer syndromes including but are not limited to:

    * Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Gardner's Syndrome
    * Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis
    * Cronkhite-Canada Syndrome, Neurofibromatosis and Familial Hyperplastic Polyposis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged 45 years or older, who are at typical average-risk of developing colorectal neoplasms and are considered enrolled after understanding and consenting to ICF. Additional subjects outside the intended us population can be enrolled onto the clinical trial but are not eligible for primary endpoint analysis.
Sampling Method: Non-Probability Sample
Enrollment: 12500 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
CRC Sensitivity | Through study completion, an average of 5 years.
  ColoSense sensitivity for subjects with colorectal cancer (CRC), which is the percentage of individuals with a diagnosis of CRC that were detected as positive by the ColoSense test.
AA Sensitivity | Through study completion, an average of 5 years.
  ColoSense sensitivity for subjects with advanced adenomas (AA), which is the percentage of individuals with a diagnosis of AA that were detected as positive by the ColoSense test.
SPL Sensitivity | Through study completion, an average of 5 years.
  ColoSense sensitivity for subjects with serrated precancerous lesions (SPL), which is the percentage of individuals with a diagnosis of SPL that were detected as positive by the ColoSense test.
NEG Specificity | Through study completion, an average of 5 years.
  ColoSense specificity for subjects with negative findings, which is the percentage of individuals with a diagnosis of negative findings that were detected as negative by the ColoSense test.

CONTACTS AND LOCATIONS:
Locations (1):
- Decentralized Study, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No